CLINICAL TRIAL: NCT01045772
Title: A Single-Centre, Open Label Study of the Safety and Tolerability of Rilonacept in Subjects Living in Germany With Muckle-Wells Syndrome (MWS), a Cryopyrin-Associated Periodic Syndrome (CAPS), or Schnitzler Syndrome (SchS)
Brief Title: Safety and Tolerability of Rilonacept in Muckle-Wells Syndrome (MWS) or Schnitzler Syndrome (SchS)
Acronym: ACCILTRA1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Karoline Krause, Karoline Krause, MD, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCILTRA1; EudraCT Number: 2006-004290-97 (Other: EMEA)
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Muckle-Wells Syndrome; Schnitzler Syndrome
Keywords: Schnitler syndrome, Muckle-Wells syndrome, anti-IL-1
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes; Schnitzler Syndrome | interventions — rilonacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IL-1 trap (Experimental)
  Interventions: Drug: rilonacept

INTERVENTIONS:
Drug: rilonacept — 160mg of rilonacept 1x/week
  Other Names: Arcalyst

SUMMARY:
This is a single-center open label study of the IL-1 transfusion protein rilonacept in subjects with Muckle-Wells syndrome (MWS), or Schnitzler syndrome (SchS) in Germany. Prospective subjects will be recruited from a patient population previously characterized in an observational study, and from referrals within the German CAPS community; SchS subjects will be recruited through the Charité Patient pool.

The Baseline phase will begin with the Screening visit (day -21 = Visit 1) and continue for three weeks; DHAFs (Daily Health Assessment Forms) will be collected from all subjects from Day - 21 to Day 0. DHAF information including MWAS (Muckle-Wells Activity Score), or SCHAS (Schnitzler Activity Score) values from this period will be used for the baseline phase evaluation. Inclusion to receive rilonacept will occur on day 0 (= Visit 2).

On day 0 eligible subjects will receive a loading dose of two subcutaneous (S.C.) injections of rilonacept for a total of 320 mg. Subsequent study drug injections of rilonacept 160 mg will be administered once a week for four weeks. After subjects complete this initial 4-week treatment phase, they will be eligible to receive rilonacept 160 mg once weekly for 48 weeks during the extended treatment phase.

DHAFs will be used to assess symptoms throughout the study. Overall a max. of 12 subjects with either MWS or SchS will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older)
* Symptomatic MWS diagnosis based on family history of MWS and evidence of a genetic mutation in CIAS1, or Symptomatic SchS
* Able to read, understand and willing to sign the informed consent form and abide with study procedures
* Able to read, understand and complete study-related questionnaires (subjects must complete their diaries for ≥ 11 of the 21 days prior to Visit 2)
* Willing, committed and able to return for all clinic visits and complete all study-related procedures, including willingness to self-administer SC injections or to have SC injections administered by a qualified person
* In females of childbearing potential: Negative pregnancy test; males and females willing to use highly effective contraception (Pearl-Index < 1).
* In men: Willingness to utilize highly effective contraception and to not have their partner[s] become pregnant during the full course of the study
* All subjects will have received a normal Chest radiograph (CXR) within 6 months prior to enrollment (signing of consent) which notes the absence of calcified granulomas and/or pleural scarring consistent with tuberculosis
* Subjects are considered eligible, if active tuberculosis is ruled out with appropriate measurements (e.g. PPD skin test, QuantiFERON-TB)

Exclusion Criteria:

* Treatment with a live (attenuated) virus vaccine during three months prior to visit 2
* Current or recent treatment (less than 5 half lives) with a TNF inhibitor
* Concurrent /ongoing treatment with Anakinra (Kineret)
* An abnormal chest radiograph consistent with clinical signs of prior or present tuberculosis infection whether or not previously treated with anti-tuberculosis agents
* A history of listeriosis, active tuberculosis, persistent chronic or active infection(s) requiring treatment with parenteral antibiotics, parenteral antivirals, or parenteral antifungals within four weeks, or oral antibiotics, oral antivirals, or oral antifungals within four weeks prior to the Screening visit
* Significant concomitant illness such as, but not limited to, cardiac, renal, neurological, endocrinological, metabolic, lymphatic or hematological disease that would adversely affect the subject's participation or evaluation in this study
* Active systemic inflammatory condition including, but not limited to, rheumatoid arthritis, systemic lupus erythematosis, polymyalgia rheumatics, vasculitis, or myositis
* History of fibromyalgia or chronic fatigue syndrome Evidence of current HIV, Hepatitis B, or Hepatitis C infection by clinical or serological history
* History of malignancies including malignant hematological disorders other than a successfully treated non-metastatic cutaneous, basal, or squamous cell carcinoma and/or in situ cervical cancer within five years of the Screening visit
* History of a demyelinating disease or multiple sclerosis
* Severe respiratory disease, including, but not limited to severe bronchiectasis, chronic obstructive pulmonary disease, bullous lung disease, uncontrolled asthma, or pulmonary fibrosis
* Known hypersensitivity to CHO cell derived therapeutics or proteins or any components of rilonacept
* Presence of any of the following laboratory abnormalities at enrollment visit: creatinine >1.5 x Upper Limit of Normal (ULN), WBC <3.6 x 103/mm3; platelet count <150,000 mm3; ALT or AST >2.0 x ULN
* Lactating females or pregnant females
* Enrollment in another investigational treatment or device study or use of an investigational agent, or no completion of less than 4 weeks or 5 half-lives, whichever is longer, since end of another investigational device or drug trial
* Subjects for whom there is concern about compliance with the protocol procedures
* Any medical condition which, in the opinion of the Investigator, would interfere with participation in the study or place the subject at risk
* Present History of substance abuse (drug or alcohol) or any other factor (e.g., serious psychiatric condition) that could limit the subject's ability to comply with study procedures
* Subjects who are detained officially or legally to an official institute
* Deafness
* Dementia due to cerebral amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability parameters (including physical examination, PPD tuberculosis skin test, review of recent chest radiograph, electrocardiograms, routine safety laboratory assessments, clinical observations, vital signs, and adverse event reporting) | 1 year

SECONDARY OUTCOMES:
Change of the mean MWAS (Muckle-Wells Activity Score) and SCHAS (Schnitzler Activity Score) from the 21-day baseline phase (day -21 to day 0) to the last 21 days of the first 4 weeks initial treatment phase (day 7 to 28) of the study. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, MD, Principal Investigator — Allergie-Centrum-Charité, Charité University Berlin, Germany
Locations (1):
- Charité University Hospital, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Krause K, Weller K, Stefaniak R, Wittkowski H, Altrichter S, Siebenhaar F, Zuberbier T, Maurer M. Efficacy and safety of the interleukin-1 antagonist rilonacept in Schnitzler syndrome: an open-label study. Allergy. 2012 Jul;67(7):943-50. doi: 10.1111/j.1398-9995.2012.02843.x. Epub 2012 May 15. PMID 22583335